CLINICAL TRIAL: NCT04089904
Title: A Phase II Trial of Neoadjuvant Pembrolizumab for Resectable Early Stage Gastroesophageal Adenocarcinoma
Brief Title: Phase II Trial of Neoadjuvant Pembrolizumab for Patients With Early Stage Gastroesophageal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0310
Record Dates: First submitted 2019-08-20; First posted 2019-09-13 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Gastric Adenocarcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARM 1 (Experimental)
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — Patients will receive 3 cycles of pembrolizumab at 200mg intravenously on day 1 of a 3 week cycle. After 3 cycles the patients will undergo surgery

SUMMARY:
To determine the pathologic complete response (pCR) rate in patients with cT1b-T2N0 GEA treated with neoadjuvant pembrolizumab followed by surgical resection.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of untreated esophageal adenocarcinoma (AC) (including Siewert type I and II esophagogastric junction AC) or gastric AC (including Siewert type III esophagogastric junction AC), with clinical stage T1b-T2, N0, and M0.
2. Patients must undergo endoscopic ultrasound (EUS), CT chest/abdomen/pelvis with IV/PO contrast (MRI abdomen/pelvis plus noncontrast chest CT is acceptable if patient has a contraindication to iodinated dye), and PET/CT to complete staging and confirm absence of metastatic disease.
3. HER2+ and HER2- patients, and all other known molecular subsets are eligible.
4. Diagnostic laparoscopy is not mandated and can be performed as clinically indicated.
5. Eligible for surgery with curative intent
6. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
8. Measurable or non-measurable disease by RECIST 1.1 will be allowed.
9. Is willing to provide tissue for correlative studies from the primary tumor lesion at baseline and at time of surgery. Is willing to provide blood and stool samples for all ordered studies.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation.
11. Have adequate organ function as defined in the following table (Table 1). Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological

    * Absolute neutrophil count (ANC) ≥1500/µL
    * Platelets ≥100 000/µL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Renal
    * Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic
    * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN Coagulation
    * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
2. Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
  3. Previous or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer for which the patient has been previously treated and the lifetime recurrence risk is less than 30%.
  4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

     Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

     Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
  5. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
  6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
  7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
  8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
  9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
  11. Has an active infection requiring systemic therapy.
  12. Has a known history of Human Immunodeficiency Virus (HIV).
  13. Has a known history of active TB (Bacillus Tuberculosis).
  14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
  15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
  17. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catenacci, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARM 1
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ARM 1
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 46.3 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: Determine the pCR rate in patients with gastroesophageal adenocarcinoma (GEA) treated with neoadjuvant pembrolizumab followed by surgery. Regression of the primary tumor will be documented by the amount of viable tumor verses the amount of fibrosis using Becker Criteria.
Time Frame: 11 weeks
Population: The study was terminated due to low accrual. Data for this outcome was not collected.
Arm/Group | ARM 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Basic Reproduction Number (R0) Resection Rate
Description: GEA patients treated with neoadjuvant pembrolizumab using proximal, distal and circumferential margins to determine the completeness of resection. The absence of tumor cells at the proximal and distal margins will be required to be classified as an R0 resection.
Time Frame: 11 weeks
Population: The study was terminated due to low accrual. Data for this outcome was not collected.
Arm/Group | ARM 1
Number analyzed (Participants) | 0

3. Secondary Outcome: Pathologic Response Grades (PRG)
Description: To determine rates of grade 1a (complete), 1b(minimal residual disease), 2 (partial response) and 3 (no response)
Time Frame: 11 weeks
Population: The study was terminated due to low accrual. Data for this outcome was not collected.
Arm/Group | ARM 1
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With GEA Taking Pembrolizumab With Treatment-related Adverse Events
Description: Evaluate the safety/tolerability patient response of pembrolizumab in patients with GEA. Number of patients with GEA taking pembrolizumab with treatment-related adverse events as assessed by CTCAE.
Time Frame: 11 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1
Number analyzed (Participants) | 3
Participants | 1

5. Secondary Outcome: Disease Free Survival Rate (DFS)
Description: DFS rate measured from the time of the first pembrolizumab dose to disease recurrence or death.
Time Frame: 11 weeks
Population: The study was terminated due to low accrual. Data for this outcome was not collected.
Arm/Group | ARM 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival Rate (OS)
Description: Overall survival rate of patients measured from the time of first pembrolizumab dose to death.
Time Frame: 11 weeks
Population: The study was terminated due to low accrual. Data for this outcome was not collected.
Arm/Group | ARM 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | ARM 1
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM 1 (N=3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Surgical (Surgical and medical procedures) | 1 — Suture leak

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT04089904/Prot_SAP_000.pdf